CLINICAL TRIAL: NCT02191423
Title: The Effect of Oxytocin on Brain Attachment and Empathy Networks, and the Association Between the Brain Response and Treatment Outcome of Brief Dyadic Psychotherapy - in Women Suffering From Postpartum Depression
Brief Title: Oxytocin and Dyadic Psychotherapy in the Treatment of Post Partum Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TASMC-14-MB-161-CTIL
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Postpartum Depression
Keywords: postpartum Depression; Diadic psychotherapy; Oxytocin; fMRI; attachment; empathy
MeSH Terms: conditions — Depression, Postpartum | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- postpartum depression (Experimental): Women suffering from postpartum depression, assessed by fMRI and then treated by dyadic psychotherapy
  1. All participants will undergo two functional brain scans at the Tel Aviv Medical Center. The two scans will take place one week apart, one scan will include administration of oxytocin (24IU) and the other will include the use of placebo (the order in which the two different treatments is applied will be random).
  2. All women in this group participate in 8-weeks of dyadic psychotherapy (DP) at the outpatient Psychiatric Department, Tel-Aviv Medical Center.
  3. A final end-of-study clinical evaluation, will be conducted at the end of 8 weeks. The evaluation will include a psychiatric evaluation, the MADRS, and a physical examination, the mother-infant interaction will be videotaped, and the YIPTA, BDI, EPDS & STAI will be administered. Salivary OXT samples will be collected from the mother and from the infant and infants will undergo a developmental assessment.
  Interventions: Drug: Oxytocin; Drug: placebo; Behavioral: Dyadic psychotherapy
- normal controls (Other): Normal control women not suffering from postpartum depression assessed by fMRI
  1. All participants will undergo two functional brain scans at the Tel Aviv Medical Center. The two scans will take place one week apart, one scan will include administration of oxytocin (24IU) and the other will include the use of placebo (the order in which the two different treatments is applied will be random).
  2. A final end-of-study clinical evaluation, will be conducted at the end of 8 weeks. The evaluation will include a psychiatric evaluation, the MADRS, and a physical examination, the mother-infant interaction will be videotaped, and the YIPTA, BDI, EPDS & STAI will be administered. Salivary OXT samples will be collected from the mother and from the infant and infants will undergo a developmental assessment.
  Interventions: Drug: Oxytocin; Drug: placebo

INTERVENTIONS:
Drug: Oxytocin — administered pre-fMRI assessment
  Other Names: Syntocinon
Drug: placebo — administered pre-fMRI assessment
Behavioral: Dyadic psychotherapy
  Arms: postpartum depression

SUMMARY:
Rationale and Hypotheses of the Current Research: the investigators speculate that mothers suffering from PPD exhibit high levels of depression and low levels of OXT, hence experiencing the interaction with their child as less rewarding, which in turn promote further depressive symptoms and interfere with child development. While dyadic psychotherapy has been studied in this context, it is unknown which depressed women will respond to this type of therapy, and whether such a response is mediated by the pro-bonding effect of oxytocin.

The aim of this study is three-fold:

1. To study the effect of the administration of a single dose (24IU) of oxytocin on cerebral circuit processing and connectivity of empathy and attachment.
2. To examine whether the clinical response of mothers suffering from postpartum depression to short term dyadic psychotherapy (based on improved mother-child interactions) can be predicted by a unique brain response pattern to oxytocin.
3. To assess the relationship between levels of oxytocin in mother and baby and the effectiveness of psychological dyadic treatment on mothers suffering from postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Women of all ages who are 3 to 8 months post-partum.
* Women who have completed a minimum of 12 years of education.
* Women who are willing and able to provide informed consent for their participation and after the study has been explained. Infant participation will be allowed after consent has been obtained from mothers.
* Current DSM-IV-TR diagnosis of PPD disorder as confirmed by SCID (administered as part of the study of protocol number PPD1, proposed to the Helsinki committee on June 2014).
* Symptoms: BDI total score >9, EPDS total score >10
* Treatment with antidepressants will be allowed provided that patients have been on the medication for at least 4 weeks prior to entry into the pre-treatment assessment phase of the study.

Exclusion Criteria:

* Unwilling or unable, in the opinion of the investigator, to comply with study instructions.
* Pregnant women.
* Clinically significant medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning).
* Women with significant risk of committing suicide or harming others in the opinion of the psychiatrist.
* Women with a current DSM-IV-TR substance or alcohol abuse. However, patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
* Women who suffers from depression due to physical condition.
* Women who suffers from severe major depression (MADRAS>30)
* Women who suffers from chronic depression (over 6 months)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Effect of the administration of oxytocin on cerebral circuit processing | Two functional brain scans one week after admission to the study (week2)
  1. This paradigm assesses empathic responses to images of individuals experiencing sad, anxious and happy events. Images are preceded by social context (i.e. "this person just won the lottery"). Control condition presents participants with images of people performing everyday actions.
  3.we generated 15 short screenplays containing triggers for both types of empathy. Each of the screenplays depicts a situation in which the characters pose a negatively-valenced bodily state (e.g. crying, itching, choking), which we expect to elicit embodied simulation in the viewer.
  2. This paradigm examines maternal FMRI responses to infant related video vignettes. Stimuli include movies of mothers' own infant vs strange infant during solitary play and mother-infant interaction.
Interactional measures-CIB | pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  The Coding Interactive Behavior Manual (CIB) (Feldman 1998), a well-validated system for coding dyadic interactions, by individuals blind to the study group that the participant is a member in. The following behaviors will be compute: Parents behavior; Child behavior; Dyadic behavior; Lead-Lag Relationship
Interactional measures-Noldus | pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  Micro-analytic coding of synchrony- on a computerized system (Noldus, The Vaggenigen, Netherlands), coded on a computerized system that allows for .01-second exactness. Consistent with previous research on parent-infant synchrony (Feldman and Eidelman, 2004, 2007). Four non-verbal categories of parenting behavior and four non-verbal categories of infant behavior will be coded and each category will include a set of mutually exclusive codes.

SECONDARY OUTCOMES:
Maternal depression symptoms measures- BDI | mothers will complete the BDI once a week during the 8-week trial, as well as in the pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  Beck Depression Inventory- BDI (Beck, Ward, Mendelson, Mock, and Erbaugh, 1961) is designed to assess the severity of depression while referring to affective, cognitive, physical and behavioral aspects.
  The BDI consists of 21 items, divided in to 3 factors: sadness / negative self perception, psycho-motor deceleration and somatic depression. Every item consists of 4 sentences for self-esteem, in a scale of 0-3, according to the degree of depression. Scores of 9 or above indicate elevated depressive symptoms and a risk for MDD (Kendall, Hollon, Beck, et al 1987). The BDI is a widely used inventory which was found to be well validated and highly coefficient (for a meta analysis see: Beck, Steer, & Garbin, 1988).
Maternal depression symptoms measures - EPDS | pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  Edinburgh Postnatal Depression Scale- EPDS, (Cox, Holden, Sagovsky, 1987) is designed in order to screen for postnatal depression in the community. The EPDS is a brief (10-item) scale. The questions focus on the psychological rather than the somatic aspects of depression and explore 2 distinct domains of negative affect: depressive symptoms (7 items) and anxiety (3 items) (Kabir, Sheeder and Kelly, 2008). Subjects respond to items on a 4 point Likert scale (of 0-3), resulting in a total score range between 0 and 30. Scores of 10 or above indicate elevated depressive symptoms and a risk for PPD (Cox, Holden, Sagovsky, 1987). The EPDS is a widely used scale which was found to be well validated and highly coefficient (Cox, Holden, Sagovsky, 1987; Kabir, Sheeder and Kelly ,2008; Murray & Carothers, 1990).
Maternal anxiety measures-STAI | mothers will complete the STAI once a week during the 8-week trial, as well as in the pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  State- Trait Anxiety Inventory- STAI (Spielberger, Gorsuch, and Lushene, 1970) assesses levels of situational and trait anxiety. The STAI contains 40 declarations, 20 of which refer to situational anxiety and 20 of which refer to trait anxiety. Subjects will indicate on a scale of 1-4 (1=not it all, 4=to a large extent) to what extent they think the declaration is accurate in their case. Trait anxiety scores of above 43 are considered a risk indicator for anxiety disorders (Spielberger, et al., 1970). The STAI is a widely used inventory which was found to be well validated and highly coefficient (Anastasi, 1988).
Physiological measures-Salivary OXT | both mothers and infants will give six saliva samples; once a other week during the 8-week trial, as well as in the pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  Salivary OXT -in order to examine OXT and reactivity curve in PPD women and their infants
Maternal thought and action measures | mothers will complete the YIPTA twice; in the pre (baseline at week 1) and post (week 11) experimental trial assessments. Data will be presented up to 1 year
  Maternal thoughts and actions will be assessed with the Yale Inventory of Parental Thoughts and Actions (YIPTA) - a semi-structured interview which provides a validated measure of parental worries, comprising a range of anxious intrusive thoughts and harm avoidant behaviors (AITHAR; Feldman, Weller, Leckman, Kuint, & Eidelman, 1999; Leckman et al., 2004; Leckman et al., 1999; Mayes, Swain, Feldman, & Leckman, 2008). Such thoughts and behaviors include concerns about the baby's physical environment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel